CLINICAL TRIAL: NCT01514734
Title: Assessing the Efficacy and Tolerability of AZARGA® (Brinzolamide 1%/Timolol 0.5% Fixed Combination) as Replacement Therapy in Patients on Brimonidine 0.2%/Timolol 0.5% Fixed Combination Therapy (COMBIGAN®) in Brazil
Brief Title: Assessing the Efficacy and Tolerability of AZARGA® (Brinzolamide 1%/Timolol 0.5% Fixed Combination) as Replacement Therapy in Patients on COMBIGAN® (Brimonidine 0.2%/Timolol 0.5% Fixed Combination) Therapy in Brazil
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-11-191
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-08

CONDITIONS: Glaucoma
Keywords: Primary open-angle glaucoma; Ocular hypertension; Pigment dispersion glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Azarga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZARGA (Experimental): Brinzolamide/timolol maleate fixed combination, one drop self-administered in study eye(s) twice a day for 8 weeks
  Interventions: Drug: Brinzolamide/timolol maleate fixed combination

INTERVENTIONS:
Drug: Brinzolamide/timolol maleate fixed combination — Commercially marketed topical ocular agent for the treatment of open-angle glaucoma (OAG) or ocular hypertension.
  Other Names: AZARGA®

SUMMARY:
The purpose of this study was to assess the efficacy and tolerability of changing to AZARGA® from prior COMBIGAN® pharmacotherapy in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Clinical diagnosis of ocular hypertension, exfoliative open-angle glaucoma, or pigment dispersion glaucoma in at least one eye (study eye).
* Be on a stable intraocular pressure (IOP) lowering regimen within 30 days of the Screening Visit.
* IOP considered safe in both eyes in such a way that should assure clinical stability of vision and optic nerve throughout the study period.
* Best corrected visual acuity of 6/60 (20/200 Snellen; 1.0 LogMAR) or better in each eye.
* IOP between 19 and 35 mmHg in at least one eye (which would be the study eye) while on brimonidine/timolol fixed combination therapy.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Presence of other primary or secondary glaucoma not listed in inclusion criteria #2.
* History of ocular herpes simplex.
* Abnormality preventing reliable applanation tonometry.
* Corneal dystrophies.
* Concurrent infectious/noninfectious conjunctivitis, keratitis, or uveitis in either eye. Blepharitis or non-clinically significant conjunctival injection is allowed.
* Intraocular conventional surgery or laser surgery in study eye(s) less than three months prior to the Screening Visit.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause.
* Use of systemic medications known to affect IOP which have not been on a stable course for 7 days prior to the Screening Visit or an anticipated change in the dosage during the course of the study.
* Pregnant or lactating.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Hubatsch, M.Sc., Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZARGA
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AZARGA
Number analyzed (Participants) | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 58.56 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  Brazil | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) at 8 Weeks From Baseline (Prior Therapy).
Description: Intraocular pressure was measured by Goldmann applanation tonometry. Data for the worse eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | AZARGA
Number analyzed (Participants) | 9
millimeters mercury (mmHg) | -0.89 (4.14)

ADVERSE EVENTS:
Arm/Group | AZARGA
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.